CLINICAL TRIAL: NCT03448159
Title: FLOW Trial: Fluoxetine to Open the Critical Period Time Window to Improve Motor Recovery After Stroke
Brief Title: Fluoxetine Opens Window to Improve Motor Recovery After Stroke
Acronym: FLOW
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: University of British Columbia (Other); Sunnybrook Health Sciences Centre (Other); University of Calgary (Other); Dalhousie University (Other); Parkwood Hospital, London, Ontario (Other); Riverview Health Centre Foundation (Other); Memorial University of Newfoundland (Other); Applied Health Research Centre (Other); Brain Canada (Other); Heart and Stroke Foundation Canadian Partnership for Stroke Recovery (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18-6002; CTO #1465 (Other: Clinical Trials Ontario)
Record Dates: First submitted 2018-02-21; First posted 2018-02-27 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Stroke; Cerebrovascular Accident; Cerebral Infarction; Brain Infarction; Brain Ischemia; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Vascular Diseases
Keywords: Stroke; Exercise; Fluoxetine; Randomized Control Trial; Rehabilitation
MeSH Terms: conditions — Stroke; Cerebral Infarction; Brain Infarction; Brain Ischemia; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Vascular Diseases; Motor Activity | interventions — Fluoxetine; Sugars; Resistance Training

STUDY DESIGN:
Intervention Model Description: Arm 1: Intervention group (will receive the trial drug, fluoxetine, as well as an exercise intervention) Arm 2: Placebo group (will receive a placebo as well as an exercise intervention
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fluoxetine Hydrochloride (Experimental): Fluoxetine (Prozac) will be administered to this group. A ramp up period of 3-5 weeks will take place where the patient takes 10mg of Prozac per day. After that, the participant will take the regular dose of 20mg for the duration of the exercise intervention (12 weeks).
  Interventions: Drug: Fluoxetine Hydrochloride; Behavioral: Exercise Program
- Placebo (Placebo Comparator): An over-encapsulated placebo, or "sugar pill" (so it appears identical to the trial drug) will be administered to this group. During the 3-5 week ramp up period for the experimental group, these participants will take a placebo identical to the 10mg Prozac capsule. After that, the participant will take a placebo identical to the 20mg Prozac capsule for the duration of the exercise intervention (12 weeks).
  Interventions: Other: Placebo; Behavioral: Exercise Program

INTERVENTIONS:
Drug: Fluoxetine Hydrochloride — Half of the participants will take fluoxetine for a period of 15-17 weeks (depending on ramp-up period).
  Other Names: Prozac
  Arms: Fluoxetine Hydrochloride
Other: Placebo — Half of the participants will take the a placebo for a period of 15-17 weeks (depending on ramp-up period).
  Other Names: "Sugar" Pill
  Arms: Placebo
Behavioral: Exercise Program — All participants will take part in a 12-week exercise program. The program will run 3 times/week, 1 hour/class.

SUMMARY:
The FLOW trial is a randomized placebo-controlled trial analyzing the effect of coupling an anti-depressant, fluoxetine (Prozac), and exercise to improve motor recovery following a stroke.

DETAILED DESCRIPTION:
FLOW Trial is a randomized, placebo-controlled, blinded phase II trial evaluating the efficacy of coupling antidepressant therapy (e.g., selective serotonin reuptake inhibitor - fluoxetine) with exercise rehabilitation across multiple Canadian sites in 176 stroke patients. 88 patients will be enrolled in each arm of the study. Both groups will receive an exercise program in addition to standard of care rehabilitation, but only one group (the intervention group) will receive the active drug fluoxetine.

Study participants will be evaluated at baseline, post-exercise program and 6-months post-exercise program. While enrolled in the study, participants will be required to take part in a 12 week, 3 times per week exercise program. Evaluators and patients will be blind to the treatment administered. The trial is constructed with randomization to remove selection and allocation biases and to ensure greater validity in observed differences in the outcome measures. The Applied Health Research Centre (AHRC) in Toronto will act as the coordinating and analysis center.

ELIGIBILITY:
Inclusion Criteria:

1. 25 years of age or older
2. Days post stroke must be between 2 to 12 months when enrolled (i.e. day of consent)
3. Patient-reported hemiparesis of the lower extremity

Exclusion Criteria:

1. Patients with subarachnoid hemorrhage
2. Pre-morbid modified Rankin score > 2
3. Substantial premorbid disability or pre-existing deficit or language comprehension deficit that could interfere with assessments
4. Diagnosis of major depressive disorder/anxiety disorder requiring antidepressant use within 6 weeks of enrolment
5. Taking neuroleptic drugs, benzodiazepines, monoamine oxidase inhibitors within 30 days of enrolment
6. Unstable serious medical condition (e.g., terminal cancer, renal or liver failure, congestive heart failure)
7. Resting blood pressure exceeding 180/100mmHg
8. Requires more than a one person assist for transfer
9. Planned surgery that would affect participation in the trial
10. Participating in another formal lower limbs exercise program more than one day per week
11. History of QT prolongation or concomitant use of clearly identified potential QT prolonging drugs, at the investigators discretion (e.g. amiodarone, bepridil, dysopyramide, dofetilide, flecainide, ibutilide, procainamide, propafenone, quinidine, sotalol, phenothiazines, pimozide, ziprasidone, TCAs, halofantrine, cisapride, and probucol)
12. History of glaucoma
13. Patients with a history of thrombocytopenia or clinically significant bleeding disorder or use of NSAID, ASA or other anticoagulants, at the investigators' discretion
14. History of convulsive disorders
15. Potential pregnancy (per screening algorithm)
16. Patients with an ongoing history of illicit drug use and/or alcohol abuse
17. Patient unwilling or unable to comply with trial requirements
18. Patient unable to understand English or communicate with the study team with staff support or translation services

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Lower Extremity Score | Following completion of the 12-week exercise intervention
  Fugl-Meyer Lower Extremity Assessment assesses motor and sensorimotor impairment in the lower extremities. Total score is between 0 and 34. Sub-scales include: proximal (0-18), knee/ankle (0-10) and coordination/speed (0-6). Higher scores indicate better performance. Sub-scale scores are summed to calculate total score.

SECONDARY OUTCOMES:
6 Minute Walk Test / 10 Meter Walk Test | Following completion of the 12-week exercise intervention and 6-months post-exercise intervention
  Physical Measurement - Ambulatory Function
Knee Strength | Following completion of the 12-week exercise intervention and 6-months post-exercise intervention
  Physical Measurement- Lower Limb Strength
Berg Balance Assessment | Following completion of the 12-week exercise intervention and 6-months post-exercise intervention
  Physical Measurement - Balance Function
Grip Strength | Following completion of the 12-week exercise intervention and 6-months post-exercise intervention
  Physical Measurement - Grip Strength
Waist-to-Hip Ratio | Following completion of the 12-week exercise intervention and 6-months post-exercise intervention
  Physical Measurement - Health Measurement
Body Mass Index | Following completion of the 12-week exercise intervention and 6-months post-exercise intervention
  Physical Measurement - Health Measurement
Stroke Impact Scale | Following completion of the 12-week exercise intervention and 6-months post-exercise intervention
  Stroke-specific, self-report, health status measure. Assesses multiple domains on a 5-point Likert scale. Domains include: strength (4-20), hand function (5-25), activities of daily living/instrumental activities of daily living (10-50), mobility (9-45), communication (7-35), emotion (9-45), memory and thinking (7-35), and participation (8-40). An extra question asks that the patient rate on a scale from 0 - 100 how much they feel that he/she has recovered from his/her stroke. The 4 physical domains (strength, hand function, mobility and activities of daily living) can be summed together to create a single, physical dimension score (28-140) while all other domains should remain separate. Higher scores indicate better function.
Fugl-Meyer Lower Extremity Score | 6-months post-exercise intervention
  Impairment Measurement (see description above)
Fugl-Meyer Upper Extremity Score | Following completion of the 12-week exercise intervention and 6-months post-exercise intervention
  Fugl-Meyer Upper Extremity Assessment assesses motor and sensorimotor impairment in the upper extremities. There is no total score for this measure. Sub-scales include: upper extremity (0-36), wrist (0-10), hand (0-14), coordination/speed (0-6) (which can be combined to form a total motor function score out of 66), and sensation (0-4). Higher scores indicate better performance.
Patient Health Questionnaire (PHQ)-9 | Following completion of the 12-week exercise intervention and 6-months post-exercise intervention
  Depression Measurement
Simple and Choice Reaction Time Test | Following completion of the 12-week exercise intervention and 6-months post-exercise intervention
  Cognitive Measurement
Trail Making Test - A & B | Following completion of the 12-week exercise intervention and 6-months post-exercise intervention
  Cognitive Measurement
Montreal Cognitive Assessment (including 5 word recall and clock test) | Following completion of the 12-week exercise intervention and 6-months post-exercise intervention
  Cognitive Measurement
Fasting Blood Draws | Following completion of the 12-week exercise intervention and 6-months post-exercise intervention
  Biological Biomarker

CONTACTS AND LOCATIONS:
Overall Officials: Mark Bayley, MD, Principal Investigator — University Health Network, Toronto; Courtney Pollock, PhD, Principal Investigator — University of British Columbia & GF Strong Rehab Centre; Bradley MacIntosh, PhD, Principal Investigator — Sunnybrook Health Sciences Centre; Sean Dukelow, MD, Principal Investigator — University of Calgary; Sepideh Pooyania, MD, Principal Investigator — Riverview Health Centre; Michelle Ploughman, PhD, Principal Investigator — Memorial University of Newfoundland; Marilyn Mackay-Lyons, PhD, Principal Investigator — Dalhousie University; Robert Teasell, MD, Principal Investigator — Parkwood Institute
Locations (8):
- Canada (8):
  - University of Calgary, Calgary, Alberta
  - University of British Columbia & GF Strong Centre, Vancouver, British Columbia
  - Riverview Health Centre, Winnipeg, Manitoba
  - Memorial University of Newfoundland, St. John's, Newfoundland and Labrador
  - Dalhousie University, Halifax, Nova Scotia
  - Parkwood Institute, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Toronto Rehabilitation Institute - University Health Network, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided
Unused blood samples will be processed and centrally stored in cryovials in a minus 80 degrees freezer for future analyses under the supervision of Study Investigator, Dr. Sandra Black (Sunnybrook, M6 West, 2075 Bayview Avenue, Toronto). The intent is to make the stored frozen cryovials available to all Heart and Stroke Foundation Canadian Partnership of Stroke Recovery (CPSR) investigators to apply for access, but it is currently undecided if other researchers will be allowed to apply for access to the samples. Access will be controlled by a Subcommittee of CPSR Investigators who will review and approve requests and oversee access to the biobank. Stored cryovials will remain at Sunnybrook under the supervision of Dr. Sandra Black for a period of up to 10 years.

REFERENCES:
- [Background] Alexander LD, Black SE, Patterson KK, Gao F, Danells CJ, McIlroy WE. Association between gait asymmetry and brain lesion location in stroke patients. Stroke. 2009 Feb;40(2):537-44. doi: 10.1161/STROKEAHA.108.527374. Epub 2008 Dec 24. PMID 19109546
- [Background] AVERT Trial Collaboration group. Efficacy and safety of very early mobilisation within 24 h of stroke onset (AVERT): a randomised controlled trial. Lancet. 2015 Jul 4;386(9988):46-55. doi: 10.1016/S0140-6736(15)60690-0. Epub 2015 Apr 16. PMID 25892679
- [Background] Salbach NM, Wood-Dauphinee S, Desrosiers J, Eng JJ, Graham ID, Jaglal SB, Korner-Bitensky N, MacKay-Lyons M, Mayo NE, Richards CL, Teasell RW, Zwarenstein M, Bayley MT; Stroke Canada Optimization of Rehabilitation By Evidence - Implementation Trial (SCORE-IT) Team. Facilitated interprofessional implementation of a physical rehabilitation guideline for stroke in inpatient settings: process evaluation of a cluster randomized trial. Implement Sci. 2017 Aug 1;12(1):100. doi: 10.1186/s13012-017-0631-7. PMID 28764752
- [Background] Bensimon K, Herrmann N, Swardfager W, Yi H, Black SE, Gao FQ, Snaiderman A, Lanctot KL. Kynurenine and depressive symptoms in a poststroke population. Neuropsychiatr Dis Treat. 2014 Sep 22;10:1827-35. doi: 10.2147/NDT.S65740. eCollection 2014. PMID 25285006
- [Background] Berends HI, Nijlant J, van Putten M, Movig KL, IJzerman MJ. Single dose of fluoxetine increases muscle activation in chronic stroke patients. Clin Neuropharmacol. 2009 Jan-Feb;32(1):1-5. PMID 19536922
- [Background] Biernaskie J, Chernenko G, Corbett D. Efficacy of rehabilitative experience declines with time after focal ischemic brain injury. J Neurosci. 2004 Feb 4;24(5):1245-54. doi: 10.1523/JNEUROSCI.3834-03.2004. PMID 14762143
- [Background] Billinger SA, Arena R, Bernhardt J, Eng JJ, Franklin BA, Johnson CM, MacKay-Lyons M, Macko RF, Mead GE, Roth EJ, Shaughnessy M, Tang A; American Heart Association Stroke Council; Council on Cardiovascular and Stroke Nursing; Council on Lifestyle and Cardiometabolic Health; Council on Epidemiology and Prevention; Council on Clinical Cardiology. Physical activity and exercise recommendations for stroke survivors: a statement for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2014 Aug;45(8):2532-53. doi: 10.1161/STR.0000000000000022. Epub 2014 May 20. PMID 24846875
- [Background] Bradbury EJ, Moon LD, Popat RJ, King VR, Bennett GS, Patel PN, Fawcett JW, McMahon SB. Chondroitinase ABC promotes functional recovery after spinal cord injury. Nature. 2002 Apr 11;416(6881):636-40. doi: 10.1038/416636a. PMID 11948352
- [Background] Breceda EY, Dromerick AW. Motor rehabilitation in stroke and traumatic brain injury: stimulating and intense. Curr Opin Neurol. 2013 Dec;26(6):595-601. doi: 10.1097/WCO.0000000000000024. PMID 24141528
- [Background] Chollet F, Tardy J, Albucher JF, Thalamas C, Berard E, Lamy C, Bejot Y, Deltour S, Jaillard A, Niclot P, Guillon B, Moulin T, Marque P, Pariente J, Arnaud C, Loubinoux I. Fluoxetine for motor recovery after acute ischaemic stroke (FLAME): a randomised placebo-controlled trial. Lancet Neurol. 2011 Feb;10(2):123-30. doi: 10.1016/S1474-4422(10)70314-8. Epub 2011 Jan 7. PMID 21216670
- [Background] Cumberland Consensus Working Group; Cheeran B, Cohen L, Dobkin B, Ford G, Greenwood R, Howard D, Husain M, Macleod M, Nudo R, Rothwell J, Rudd A, Teo J, Ward N, Wolf S. The future of restorative neurosciences in stroke: driving the translational research pipeline from basic science to rehabilitation of people after stroke. Neurorehabil Neural Repair. 2009 Feb;23(2):97-107. doi: 10.1177/1545968308326636. PMID 19189939
- [Background] Dhami KS, Churchward MA, Baker GB, Todd KG. Fluoxetine and citalopram decrease microglial release of glutamate and D-serine to promote cortical neuronal viability following ischemic insult. Mol Cell Neurosci. 2013 Sep;56:365-74. doi: 10.1016/j.mcn.2013.07.006. Epub 2013 Jul 19. PMID 23876875
- [Background] Dromerick AW, Edwardson MA, Edwards DF, Giannetti ML, Barth J, Brady KP, Chan E, Tan MT, Tamboli I, Chia R, Orquiza M, Padilla RM, Cheema AK, Mapstone ME, Fiandaca MS, Federoff HJ, Newport EL. Critical periods after stroke study: translating animal stroke recovery experiments into a clinical trial. Front Hum Neurosci. 2015 Apr 29;9:231. doi: 10.3389/fnhum.2015.00231. eCollection 2015. PMID 25972803
- [Background] Espinera AR, Ogle ME, Gu X, Wei L. Citalopram enhances neurovascular regeneration and sensorimotor functional recovery after ischemic stroke in mice. Neuroscience. 2013 Sep 5;247:1-11. doi: 10.1016/j.neuroscience.2013.04.011. Epub 2013 Apr 13. PMID 23590907
- [Background] Goyal M, Demchuk AM, Menon BK, Eesa M, Rempel JL, Thornton J, Roy D, Jovin TG, Willinsky RA, Sapkota BL, Dowlatshahi D, Frei DF, Kamal NR, Montanera WJ, Poppe AY, Ryckborst KJ, Silver FL, Shuaib A, Tampieri D, Williams D, Bang OY, Baxter BW, Burns PA, Choe H, Heo JH, Holmstedt CA, Jankowitz B, Kelly M, Linares G, Mandzia JL, Shankar J, Sohn SI, Swartz RH, Barber PA, Coutts SB, Smith EE, Morrish WF, Weill A, Subramaniam S, Mitha AP, Wong JH, Lowerison MW, Sajobi TT, Hill MD; ESCAPE Trial Investigators. Randomized assessment of rapid endovascular treatment of ischemic stroke. N Engl J Med. 2015 Mar 12;372(11):1019-30. doi: 10.1056/NEJMoa1414905. Epub 2015 Feb 11. PMID 25671798
- [Background] Hachinski V, Iadecola C, Petersen RC, Breteler MM, Nyenhuis DL, Black SE, Powers WJ, DeCarli C, Merino JG, Kalaria RN, Vinters HV, Holtzman DM, Rosenberg GA, Wallin A, Dichgans M, Marler JR, Leblanc GG. National Institute of Neurological Disorders and Stroke-Canadian Stroke Network vascular cognitive impairment harmonization standards. Stroke. 2006 Sep;37(9):2220-41. doi: 10.1161/01.STR.0000237236.88823.47. Epub 2006 Aug 17. PMID 16917086
- [Background] Hackett ML, Duncan JR, Anderson CS, Broad JB, Bonita R. Health-related quality of life among long-term survivors of stroke : results from the Auckland Stroke Study, 1991-1992. Stroke. 2000 Feb;31(2):440-7. doi: 10.1161/01.str.31.2.440. PMID 10657420
- [Background] Harris JE, Eng JJ, Miller WC, Dawson AS. A self-administered Graded Repetitive Arm Supplementary Program (GRASP) improves arm function during inpatient stroke rehabilitation: a multi-site randomized controlled trial. Stroke. 2009 Jun;40(6):2123-8. doi: 10.1161/STROKEAHA.108.544585. Epub 2009 Apr 9. PMID 19359633
- [Background] Hsieh YW, Wang CH, Sheu CF, Hsueh IP, Hsieh CL. Estimating the minimal clinically important difference of the Stroke Rehabilitation Assessment of Movement measure. Neurorehabil Neural Repair. 2008 Nov-Dec;22(6):723-7. doi: 10.1177/1545968308316385. Epub 2008 Sep 5. PMID 18776067
- [Background] Hsueh IP, Hsu MJ, Sheu CF, Lee S, Hsieh CL, Lin JH. Psychometric comparisons of 2 versions of the Fugl-Meyer Motor Scale and 2 versions of the Stroke Rehabilitation Assessment of Movement. Neurorehabil Neural Repair. 2008 Nov-Dec;22(6):737-44. doi: 10.1177/1545968308315999. Epub 2008 Jul 21. PMID 18645189
- [Background] Iadecola C, Anrather J. Stroke research at a crossroad: asking the brain for directions. Nat Neurosci. 2011 Oct 26;14(11):1363-8. doi: 10.1038/nn.2953. PMID 22030546
- [Background] Jorgensen HS, Nakayama H, Raaschou HO, Vive-Larsen J, Stoier M, Olsen TS. Outcome and time course of recovery in stroke. Part I: Outcome. The Copenhagen Stroke Study. Arch Phys Med Rehabil. 1995 May;76(5):399-405. doi: 10.1016/s0003-9993(95)80567-2. PMID 7741608
- [Background] Kobayashi K, Ikeda Y, Sakai A, Yamasaki N, Haneda E, Miyakawa T, Suzuki H. Reversal of hippocampal neuronal maturation by serotonergic antidepressants. Proc Natl Acad Sci U S A. 2010 May 4;107(18):8434-9. doi: 10.1073/pnas.0912690107. Epub 2010 Apr 19. PMID 20404165
- [Background] Krakauer JW, Carmichael ST, Corbett D, Wittenberg GF. Getting neurorehabilitation right: what can be learned from animal models? Neurorehabil Neural Repair. 2012 Oct;26(8):923-31. doi: 10.1177/1545968312440745. Epub 2012 Mar 30. PMID 22466792
- [Background] Kwah LK, Harvey LA, Diong J, Herbert RD. Models containing age and NIHSS predict recovery of ambulation and upper limb function six months after stroke: an observational study. J Physiother. 2013 Sep;59(3):189-97. doi: 10.1016/S1836-9553(13)70183-8. PMID 23896334
- [Background] Langdon KD, Corbett D. Improved working memory following novel combinations of physical and cognitive activity. Neurorehabil Neural Repair. 2012 Jun;26(5):523-32. doi: 10.1177/1545968311425919. Epub 2011 Dec 9. PMID 22157145
- [Background] Levine B, Schweizer TA, O'Connor C, Turner G, Gillingham S, Stuss DT, Manly T, Robertson IH. Rehabilitation of executive functioning in patients with frontal lobe brain damage with goal management training. Front Hum Neurosci. 2011 Feb 17;5:9. doi: 10.3389/fnhum.2011.00009. eCollection 2011. PMID 21369362
- [Background] Lynch E, Hillier S, Cadilhac D. When should physical rehabilitation commence after stroke: a systematic review. Int J Stroke. 2014 Jun;9(4):468-78. doi: 10.1111/ijs.12262. Epub 2014 Mar 18. PMID 24636633
- [Background] Mackay-Lyons M, McDonald A, Matheson J, Eskes G, Klus MA. Dual effects of body-weight supported treadmill training on cardiovascular fitness and walking ability early after stroke: a randomized controlled trial. Neurorehabil Neural Repair. 2013 Sep;27(7):644-53. doi: 10.1177/1545968313484809. Epub 2013 Apr 18. PMID 23599221
- [Background] Mansfield A, Wong JS, Bryce J, Brunton K, Inness EL, Knorr S, Jones S, Taati B, McIlroy WE. Use of Accelerometer-Based Feedback of Walking Activity for Appraising Progress With Walking-Related Goals in Inpatient Stroke Rehabilitation: A Randomized Controlled Trial. Neurorehabil Neural Repair. 2015 Oct;29(9):847-57. doi: 10.1177/1545968314567968. Epub 2015 Jan 20. PMID 25605632
- [Background] Maya Vetencourt JF, Sale A, Viegi A, Baroncelli L, De Pasquale R, O'Leary OF, Castren E, Maffei L. The antidepressant fluoxetine restores plasticity in the adult visual cortex. Science. 2008 Apr 18;320(5874):385-8. doi: 10.1126/science.1150516. PMID 18420937
- [Background] McEwen D, Taillon-Hobson A, Bilodeau M, Sveistrup H, Finestone H. Virtual reality exercise improves mobility after stroke: an inpatient randomized controlled trial. Stroke. 2014 Jun;45(6):1853-5. doi: 10.1161/STROKEAHA.114.005362. Epub 2014 Apr 24. PMID 24763929
- [Background] McIntyre A, Richardson M, Janzen S, Hussein N, Teasell R. The evolution of stroke rehabilitation randomized controlled trials. Int J Stroke. 2014 Aug;9(6):789-92. doi: 10.1111/ijs.12272. Epub 2014 Mar 13. PMID 24621406
- [Background] Murphy TH, Corbett D. Plasticity during stroke recovery: from synapse to behaviour. Nat Rev Neurosci. 2009 Dec;10(12):861-72. doi: 10.1038/nrn2735. Epub 2009 Nov 4. PMID 19888284
- [Background] Nadeau SE, Wu SS, Dobkin BH, Azen SP, Rose DK, Tilson JK, Cen SY, Duncan PW; LEAPS Investigative Team. Effects of task-specific and impairment-based training compared with usual care on functional walking ability after inpatient stroke rehabilitation: LEAPS Trial. Neurorehabil Neural Repair. 2013 May;27(4):370-80. doi: 10.1177/1545968313481284. Epub 2013 Mar 15. PMID 23504552
- [Background] Pizzorusso T, Medini P, Berardi N, Chierzi S, Fawcett JW, Maffei L. Reactivation of ocular dominance plasticity in the adult visual cortex. Science. 2002 Nov 8;298(5596):1248-51. doi: 10.1126/science.1072699. PMID 12424383
- [Background] Ploughman M, Granter-Button S, Chernenko G, Tucker BA, Mearow KM, Corbett D. Endurance exercise regimens induce differential effects on brain-derived neurotrophic factor, synapsin-I and insulin-like growth factor I after focal ischemia. Neuroscience. 2005;136(4):991-1001. doi: 10.1016/j.neuroscience.2005.08.037. Epub 2005 Oct 3. PMID 16203102
- [Background] Ploughman M, Windle V, MacLellan CL, White N, Dore JJ, Corbett D. Brain-derived neurotrophic factor contributes to recovery of skilled reaching after focal ischemia in rats. Stroke. 2009 Apr;40(4):1490-5. doi: 10.1161/STROKEAHA.108.531806. Epub 2009 Jan 22. PMID 19164786
- [Background] Pollock A, St George B, Fenton M, Firkins L. Top 10 research priorities relating to life after stroke--consensus from stroke survivors, caregivers, and health professionals. Int J Stroke. 2014 Apr;9(3):313-20. doi: 10.1111/j.1747-4949.2012.00942.x. Epub 2012 Dec 11. PMID 23227818
- [Background] Portelli R, Lowe D, Irwin P, Pearson M, Rudd AG; Intercollegiate Stroke Working Party. Institutionalization after stroke. Clin Rehabil. 2005 Jan;19(1):97-108. doi: 10.1191/0269215505cr822oa. PMID 15704514
- [Background] Savitz SI, Cramer SC, Wechsler L; STEPS 3 Consortium. Stem cells as an emerging paradigm in stroke 3: enhancing the development of clinical trials. Stroke. 2014 Feb;45(2):634-9. doi: 10.1161/STROKEAHA.113.003379. Epub 2013 Dec 24. No abstract available. PMID 24368562
- [Background] Scali M, Begenisic T, Mainardi M, Milanese M, Bonifacino T, Bonanno G, Sale A, Maffei L. Fluoxetine treatment promotes functional recovery in a rat model of cervical spinal cord injury. Sci Rep. 2013;3:2217. doi: 10.1038/srep02217. PMID 23860568
- [Background] Soleman S, Yip PK, Duricki DA, Moon LD. Delayed treatment with chondroitinase ABC promotes sensorimotor recovery and plasticity after stroke in aged rats. Brain. 2012 Apr;135(Pt 4):1210-23. doi: 10.1093/brain/aws027. Epub 2012 Mar 6. PMID 22396394
- [Background] Stinear CM, Byblow WD. Predicting and accelerating motor recovery after stroke. Curr Opin Neurol. 2014 Dec;27(6):624-30. doi: 10.1097/WCO.0000000000000153. PMID 25364953
- [Background] Van Breukelen GJ. ANCOVA versus change from baseline: more power in randomized studies, more bias in nonrandomized studies [corrected]. J Clin Epidemiol. 2006 Sep;59(9):920-5. doi: 10.1016/j.jclinepi.2006.02.007. Epub 2006 Jun 23. PMID 16895814
- [Background] Vickers AJ. Analysis of variance is easily misapplied in the analysis of randomized trials: a critique and discussion of alternative statistical approaches. Psychosom Med. 2005 Jul-Aug;67(4):652-5. doi: 10.1097/01.psy.0000172624.52957.a8. PMID 16046383
- [Background] Wade DT, Skilbeck CE, Wood VA, Langton Hewer R. Long-term survival after stroke. Age Ageing. 1984 Mar;13(2):76-82. doi: 10.1093/ageing/13.2.76. PMID 6731168
- [Background] Wahl AS, Omlor W, Rubio JC, Chen JL, Zheng H, Schroter A, Gullo M, Weinmann O, Kobayashi K, Helmchen F, Ommer B, Schwab ME. Neuronal repair. Asynchronous therapy restores motor control by rewiring of the rat corticospinal tract after stroke. Science. 2014 Jun 13;344(6189):1250-5. doi: 10.1126/science.1253050. PMID 24926013
- [Background] Wang CH, Hsieh CL, Dai MH, Chen CH, Lai YF. Inter-rater reliability and validity of the stroke rehabilitation assessment of movement (stream) instrument. J Rehabil Med. 2002 Jan;34(1):20-4. doi: 10.1080/165019702317242668. PMID 11900258
- [Background] Wang D, Fawcett J. The perineuronal net and the control of CNS plasticity. Cell Tissue Res. 2012 Jul;349(1):147-60. doi: 10.1007/s00441-012-1375-y. Epub 2012 Mar 23. PMID 22437874
- [Background] Zittel S, Weiller C, Liepert J. Citalopram improves dexterity in chronic stroke patients. Neurorehabil Neural Repair. 2008 May-Jun;22(3):311-4. doi: 10.1177/1545968307312173. Epub 2008 Jan 24. PMID 18219053
- See also: Research breakthrough to revolutionize stroke treatment — http://www.heartandstroke.ca/articles/research-breakthrough-to-revolutionize-stroke-treatment
- See also: Tracking Heart Disease and Stroke in Canada — http://www.phac-aspc.gc.ca/publicat/2009/cvd-avc/pdf/cvd-avs-2009-eng.pdf